CLINICAL TRIAL: NCT01919372
Title: Intensificación y monitorización telemática Personalizada de la modificación Del Estilo de Vida en el Tratamiento de la Obesidad y la prevención Del Riesgo cardiometabólico
Brief Title: Individualized Telemedical Assistance for Lifestyle Modification in the Treatment of Obesity and Cardiometabolic Risk Prevention
Acronym: PREDIRCAM 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Grupo de Bioingenieria y Telemedicina -ETSI Telecomunicacion. Universidad Politecnica de Madrid (Unknown); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-MTP-2012-74
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Obesity Type I and II
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional assistance (Active Comparator): Usual treatment of obesity in terms of monitoring lifestyle habits
  Interventions: Other: Standard care
- Telemedic assistance (Experimental): telemedical assistance with a technological system to provide a continuous monitoring of lifestyle habits and individualized treatment of obesity
  Interventions: Device: Telemedic assistance with a technological system

INTERVENTIONS:
Device: Telemedic assistance with a technological system
  Other Names: PREDIRCAM
  Arms: Telemedic assistance
Other: Standard care
  Arms: Conventional assistance

SUMMARY:
This project is based on the contribution that could offer a technological system for a continuous monitoring, individualized treatment of obesity and prevention of cardiometabolic complications in high risk population.

The main objective of PREDIRCAM study is to evaluate the benefits obtained with the use in high cardiometabolic risk individuals of a telemedical platform integrating applications for monitoring and providing recommendations to improve lifestyle habits (diet and physical activity) in a healthier way.

The study population are obese subjects (type I or II) aged between 25 and 65 years with a 12 month follow-up. In this population it will be analysed the cost-effectiveness of a telemedic assistance with a technological system and its ability to modify lifestyle habits, reduce weight and cardiovascular risk associated parameters.

Previously to the clinical implementation, a pilot study for testing the telemedical system will be made. Efficacy and security variables will be evaluated along the study.

ELIGIBILITY:
Inclusion Criteria:

Preclinical Phase:

1. People over 18 years with or without obesity and with ability for technology management

Clinical Phase:

1. People between 18 and 65 years.
2. Obesity defined as a body mass index (BMI) greater than or equal to 30 kg/m2:

   1. Grade I or II without sleep apnea syndrome and ischemic heart disease
   2. Absence of metabolic processes (dyslipidemia) or associated hypertension requiring drug treatment at the time of inclusion in the study.
3. People with ability for technology management

Exclusion Criteria:

Preclinical Phase:

1. Serious illness and / or disabling

Clinical Phase:

1. Diabetes defining according to American Diabetes Association (ADA) criteria.
2. Subjects with moderate to severe active disease at the time of inclusion in the study protocol
3. Impaired glucose metabolism related diseases associated with diabetes mellitus or drugs interfering carbohydrate metabolism.
4. Cardiovascular disease
5. Dyslipidemia or hypertension requiring drug treatment.
6. Alcohol consumption
7. Pregnancy
8. Serious illness and / or disabling

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Weight loss | 1 year

SECONDARY OUTCOMES:
Cardiometabolic risk prevention | 1 year
  We will measure different parameters related to cardiovascular risk, such as adiponectine, tumour necrosis factor, Homeostasis Model Assessment, etc.at the beginning and at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain